CLINICAL TRIAL: NCT02160418
Title: Incentives for Daily Tooth Brushing to Reduce Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 819853
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-04

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): 36 Participants will be sent a new toothbrush and will be asked to use it in place of their current brush. They also receive twice daily reminders via sms to brush their teeth.
- Financial Incentives (Experimental): 36 Participants will receive a toothbrush and twice daily reminders to brush their teeth. They will also be offered financial incentives twice a day to brush their teeth.
  Interventions: Behavioral: Financial Incentives
- Cognitive Incentives (Experimental): 36 Participants will receive a toothbrush and twice daily reminders to brush their teeth. Twice a week, they will receive text messages (SMS) with a short quiz question related to oral hygiene behavior and oral health. Participants will receive a reward if they answer correctly via text message.
  Interventions: Behavioral: Cognitive Incentives
- Financial and Cognitive Incentives (Experimental): 36 Participants will receive a toothbrush and twice daily reminders to brush their teeth. Twice daily they receive financial incentives to brush their teeth. Twice a week, they will receive text messages (SMS) with a short quiz question related to oral hygiene behavior and oral health. Participants will receive a reward if they answer correctly via text message.
  Interventions: Behavioral: Financial and Cognitive Incentives

INTERVENTIONS:
Behavioral: Financial Incentives
  Arms: Financial Incentives
Behavioral: Cognitive Incentives
  Arms: Cognitive Incentives
Behavioral: Financial and Cognitive Incentives
  Arms: Financial and Cognitive Incentives

SUMMARY:
In this randomized controlled study, the investigators compare two classes of behavioral approaches to change habits and health outcomes with an application to dental health: cognitive vs. behavioral financial incentives. Under cognitive incentives subjects are paid to correctly answer health-related quizzes. Under behavioral incentives subjects earn money for making healthy choices. The investigators apply these incentives to toothbrushing, a daily health-related behavior critical to the prevention of dental caries and periodontal disease, two high-burden conditions among US adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 18 years, with at least 10 teeth present.

Exclusion Criteria:

* Pregnancy, uncontrolled diabetes, systemic antibiotics taken within the previous 2 months, need for referral for periodontal treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04-14 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Follow-up Gingival Index | 6 months

SECONDARY OUTCOMES:
Frequency and duration of toothbrushing | 3 months
End of treatment Gingival Index | 3 months
  Gingival Index at the end of behavioral incentives

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States